CLINICAL TRIAL: NCT03346642
Title: Combined Chemotherapy and PD-1 Antibody(SHR-1210) With or Without Low-dose Decitabine Priming for Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL):Two Stage, Phase I/II Trail
Brief Title: Two Stage Study of Combination of Chemotherapy, SHR-1210 and/or Decitabine for Relapsed/Refractory PMBCLs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-025
Record Dates: First submitted 2017-10-07; First posted 2017-11-17 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Primary Mediastinal Large B-cell Lymphoma
Keywords: Relapsed/Refractory; primary mediastinal large B-cell lymphoma; PD-1 antibody; Decitabine; GVD chemotherapy
MeSH Terms: conditions — Recurrence | interventions — Decitabine; camrelizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GVD and SHR-1210 with or without Decitabine (Experimental): This is a two stage study. For the first stage, the participants will receive the combination of GVD chemotherapy and PD-1 antibody SHR-1210. The patients enrolled into the second stage will received the combination of GVD and SHR-1210 with low-dose decitabine primed.
  Interventions: Drug: Decitabine; Drug: GVD chemotherapy; Drug: SHR-1210

INTERVENTIONS:
Drug: Decitabine — Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1 (DNMT1), which can increase tumor antigens and histocompatibility leukocyte antigen (HLA) expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function.
Drug: GVD chemotherapy — GVD regimen is a chemotherapy regimen consisted by Gemcitabine, Vinorelbine and Doxorubicine. Patients will be administrated with Gemcitabine 0.8 g/m2, Vinorelbine 30mg and Doxorubicin 20mg/m2 intravenously infusion.
Drug: SHR-1210 — SHR-1210 is a humanized anti-PD-1 monoclonal antibody.
  Other Names: PD-1 antibody, PD-1 inhibitor

SUMMARY:
This is a two stage, Phase I/II clinical trial for patients with relapsed or refractory primary mediastinal large B-cell lymphoma (rrPMBCL). In the first stage, the participants will receive GVD (Gemcitabine, Vinorelbine and Doxorubicine) chemotherapy and PD-1 antibody (SHR-1210) treatment. The safety and efficacy of combined regimen will be evaluated. If deemed safe and efficacious, the investigators will proceed to the second stage of the study. In the second stage, the participants will receive GVD chemotherapy and SHR-1210 treatment with low-dose Decitabine priming. The safety and feasibility of combined regimens will be evaluated in phase I study. The feasibility will be accessed.

ELIGIBILITY:
Inclusion Criteria:

1. All patients had histologically proven PMBCL, and Radiographically measureable disease.
2. Eastern Cooperative Oncology Group performance status 0-2
3. Disease recurring within 6 months after first-line chemotherapy or disease progression while receiving or persistent disease after first-line chemotherapy
4. Bulky disease was defined as the presence of a mediastinal mass > 4.5 cm in axial diameter or extranodal lesion > 3 cm.
5. Subjects must have received at least two prior chemotherapy regimen, and must be off therapy for at least 4 weeks prior to Day 1. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months. Subjects with Anti-PD-1 antibody are eligible which must be resistance.
6. Adequate organ function.
7. Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.
8. Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Known clinically active central nervous system involvement.
2. Any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
3. Serious uncontrolled medical disorders or active infections, pulmonary infection especially
4. Prior organ allograft.
5. Receiving any other form of immunosuppressive medication, except steroid.
6. Allogeneic hematopoietic stem cell transplantation within the last 5 years. 6） Known human immunodeficiency virus (HIV). 7） Has received a live vaccine within 30 days prior to first dose of study drug.

8） Women who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment-related adverse events (AEs) | Up to 120 days after last administration of SHR-1210
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v4.03.
Objective response rate (ORR) | Enrolled patients will be followed until death, withdrawal from study, or until 2 years.
  The antitumor efficacy of the combination treatments as measured by ORR was determined using the International Working Group 2007 criteria for malignant lymphoma (J Clin Oncol. 2007 Feb 10;25(5):579-586). Clinical response of progressive disease (PD), stable disease (SD), partial remission (PR), or complete remission (CR) will be determined at each assessment. ORR is defined as the sum of CR and PR.

SECONDARY OUTCOMES:
Complete response (CR) rate | Up to 2 years after completion of study treatment
  The CR rate will be estimated as the proportion of patients with response, with a 95% exact confidence interval.
Median progression-free survival (PFS) time | Patients will be followed until disease progression, death, withdrawal from study, or until 2 years.
  PFS time was measured from study entry to the first documentation of disease progression or death. Disease progression was determined using the International Working Group 2007 criteria for malignant lymphoma.
Median overall survival (OS) time | Patients will be followed until death, withdrawal from study, or until 2 years.
  OS time was measured from the study entry to the date of death.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Biotherapeutic Department and Pediatrics Department of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality